CLINICAL TRIAL: NCT02552420
Title: The Clinical Application of Infrared Thermal Imaging Detecting Venous Thromboembolism
Status: Completed | Type: Observational
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Fangge Deng, Principal Investigator, The First Affiliated Hospital of Guangzhou Medical University
Other Study IDs: GIRD
Record Dates: First submitted 2015-07-28; First posted 2015-09-17 (Estimated); Last update posted 2015-09-17 (Estimated); Status verified 2015-09

CONDITIONS: Deep Venous Thrombosis
Keywords: infrared thermal imaging; deep venous thrombosis
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine the effectiveness of infrared thermal imaging in adjunctive diagnostic screening for lower limb deep venous thrombosis (DVT).

ELIGIBILITY:
Inclusion Criteria:

1. Willing to participate in the trial and sign the informed consent form,
2. Aged: 18-75 years. They had been definitively diagnosed with venous thromboembolism,
3. The bed-rest immobilization time should be more than 72 hours,
4. Planing to gynecology operation,
5. The D dimer should be more than500 g • L-1,
6. There is no obvious symptoms of systemic infection two weeks before the test,
7. There is no trauma, infection, biopsy or puncture, hemorrhage and tumor in the corresponding detection site (chest and lower limbs),
8. There is no skin disease, heart, liver, kidney, gastrointestinal tract, hematopoietic system and mental, neurological has no serious diseases.

Exclusion Criteria:

1. Patients can not be good partners,
2. Doctors believe that there is any inappropriate situations.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: DVT patients included in this study had been definitively diagnosed as having DVT with CPUS and/or angiography. Included non-DVT volunteers were confirmed to be without DVT with CPUS. The healthy volunteer group matched the DVT group in number, age, and gender.
Sampling Method: Non-Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2007-09; Primary Completion 2012-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Using the Infrared Thermal Imaging to detecting Venous Thromboembolism | up to 24 months
  ① Different levels of pseudocode (white, red, pink, yellow, green, blue, black) representing related IRTI that corresponds to a color scale bar of low to high temperatures, so we can know disease's position, extent and severity by comparing with the difference of color distribution and shape in the thermal imaging.
  ②The intensity of thermal distribution is higher than normals (great than or equal 0.5 Celsius degree is unnoraml), the symmetry of thermal range is relatively increased (pixels over 0.5 ~ 1.0-fold), the difference of spatial distribution of the thermal field and the difference of statistically analyze are related to the disease.